CLINICAL TRIAL: NCT01676688
Title: Safety Study of Alfalastin (Human Alpha-1 Antitrypsin, 33.33 mg/ml) Administered at Home to Patients Suffering From Severe Forms of Primary Deficiency in Alpha-1 Antitrypsin, Phenotype PIZZ or PISZ, With Pulmonary Emphysema.
Brief Title: Safety Study of Alfalastin (Human Alpha-1 Antitrypsin) Administered at Home
Status: Completed | Type: Observational
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Other Study IDs: AlfaDom
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: alpha-1 antitrypsin; deficiency; Alfalastin; safety
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect safety data on ALFALASTIN® infusions performed at home or in out-of hospital locations.

DETAILED DESCRIPTION:
Non interventional, observational, longitudinal, prospective, multicenter, non comparative study.

ELIGIBILITY:
Participation Criteria:

* Patients above 18 y.o,
* suffering from severe forms of primary alpha-1 antitrypsin deficiency, phenotype PiZZ or PiSZ with pulmonary emphysema,
* currently treated as per routine practice, once a week, by ALFALASTIN® at home or in out-of-hospital location
* and having signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 18 y.o, suffering from severe forms of primary alpha-1 antitrypsin deficiency, phenotype PiZZ or PiSZ with pulmonary emphysema, currently treated , once a week, as per routine practice by ALFALASTIN® at home or in out-of-hospital location.
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cuvelier Antoine, Prof., Study Director — Pneumology - CHU Rouen, France; Mornex Jean-François, Prof, Study Chair — Pneumology - CHU Lyon, France; Thabut Gabriel, MD, Study Chair — Pneumology - Hôpital Bichat Paris, France